CLINICAL TRIAL: NCT05461092
Title: Regional Nerve Blocks to Improve Analgesia and Recovery in Older Adults Undergoing Spinal Fusion
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Catherine R. Olinger, Clinical Assistant Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202305284
Record Dates: First submitted 2022-06-20; First posted 2022-07-15 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Delirium; Pain, Back; Spinal Fusion; Thoracolumbar Interfascial Plane Block
MeSH Terms: conditions — Delirium; Back Pain | interventions — Hematologic Tests; Patient Health Questionnaire; Weights and Measures; Interviews as Topic

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Both patient (participant) and surgeon will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care Anesthesia without Thoracolumbar Interfascial Plane (TLIP) Block of bupivicaine. (Active Comparator): Subjects will receive standard of care anesthesia without TLIP Block of bupivicaine.
  Interventions: Diagnostic Test: Blood Test; Other: 3D CAM Delirium Severity Scoring; Other: Generalized Anxiety Disorder 7-item (GAD-7) scale; Other: Numerical Rating Score (NRS); Other: PROMIS-Pain Interference; Other: Oswestry Disability Index (ODI); Other: Saint Louis University Mental Status Examination (SLUMs); Other: Delirium Rating Scale-Revised-98 (DRS); Other: Telephone Interview for Cognitive Status - Modified (TICS-M); Other: Opioid Equivalents measured by Morphine Milligram Equivalents (MME); Other: Patient Health Questionnaire depression scale (PHQ-8); Other: Pain Catastrophizing; Other: Fear Avoidance Beliefs Questionnaire (FABQ); Other: Opioid Side Effects and Likeability Questionnaire; Other: Daily Pain Trajectory; Other: Tampa Scale of Kinesiophobia; Other: Quality of Recovery 15
- Standard of Care Anesthesia with Thoracolumbar Interfascial Plane (TLIP) Block of bupivacaine (Experimental): Patient receives standard of care anesthesia with TLIP Block of bupivacaine (local anesthetic) intraoperatively after anesthesia administration and before spinal fusion.
  Interventions: Drug: Thoracolumbar Interfascial Plane (TLIP) Block of bupivacaine; Diagnostic Test: Blood Test; Other: 3D CAM Delirium Severity Scoring; Other: Generalized Anxiety Disorder 7-item (GAD-7) scale; Other: Numerical Rating Score (NRS); Other: PROMIS-Pain Interference; Other: Oswestry Disability Index (ODI); Other: Saint Louis University Mental Status Examination (SLUMs); Other: Delirium Rating Scale-Revised-98 (DRS); Other: Telephone Interview for Cognitive Status - Modified (TICS-M); Other: Opioid Equivalents measured by Morphine Milligram Equivalents (MME); Other: Patient Health Questionnaire depression scale (PHQ-8); Other: Pain Catastrophizing; Other: Fear Avoidance Beliefs Questionnaire (FABQ); Other: Opioid Side Effects and Likeability Questionnaire; Other: Daily Pain Trajectory; Other: Tampa Scale of Kinesiophobia; Other: Quality of Recovery 15

INTERVENTIONS:
Drug: Thoracolumbar Interfascial Plane (TLIP) Block of bupivacaine — Patient receives standard of care anesthesia with TLIP Block of bupivicaine (local anesthetic) intraoperatively after anesthesia administration and before spinal fusion.
  Arms: Standard of Care Anesthesia with Thoracolumbar Interfascial Plane (TLIP) Block of bupivacaine
Diagnostic Test: Blood Test — Blood Tests measuring inflammatory markers: IL-10, MCP-1, IL-8, IL-6, TNFa
Other: 3D CAM Delirium Severity Scoring — Questionnaire that will rate each symptom of delirium
Other: Generalized Anxiety Disorder 7-item (GAD-7) scale — Questionnaire for screening and severity measurement of generalized anxiety disorder.
Other: Numerical Rating Score (NRS) — Questionnaire assessing pain intensity
Other: PROMIS-Pain Interference — Questionnaire measuring the effect of pain on patient physical, emotional, and social functioning.
Other: Oswestry Disability Index (ODI) — Questionnaire assessing disability and quality of life impairment in adults with lower back pain.
Other: Saint Louis University Mental Status Examination (SLUMs) — Questionnaire assessing baseline cognition.
Other: Delirium Rating Scale-Revised-98 (DRS) — 16 item clinician rated scale assessing delirium severity.
Other: Telephone Interview for Cognitive Status - Modified (TICS-M) — Telephone interview questionnaire evaluating patient cognitive status.
Other: Opioid Equivalents measured by Morphine Milligram Equivalents (MME) — The amount of opioids administered will be collected through patient self-report
Other: Patient Health Questionnaire depression scale (PHQ-8) — Questionnaire used to diagnose and determine the severity measure for depressive disorders.
Other: Pain Catastrophizing — Scale used to determine pain catastrophizing and it's severity.
Other: Fear Avoidance Beliefs Questionnaire (FABQ) — Questionnaire used to help predict patients that have a high pain avoidance behavior.
Other: Opioid Side Effects and Likeability Questionnaire — Survey determining adverse events related to opioid side effects and complications.
Other: Daily Pain Trajectory — Questionnaire assessing pain location, severity, impact to quality of life, and medications used to alleviate.
Other: Tampa Scale of Kinesiophobia — Questionnaire assessing Kinesiophobia
Other: Quality of Recovery 15 — Questionnaire assessing postoperative quality of recovery

SUMMARY:
This initial study is a feasibility study for implementing thoracolumbar interfascial plane, or TLIP, blocks in older adults undergoing spinal fusion. TLIP blocks are done by using anesthesia. In this case, it will be done to either side of the back where surgery will be performed. This has been shown to decrease pain the patients have post-operatively in previous research. In this study, the investigators will examine recruitment rates, completion of assessments, dropout rate, gather patient feedback, and identify barriers to performing TLIP. Further, this feasibility study will provide data to determine adequate sample size and refine methods and outcomes for a future randomized clinical trial. The ultimate goal is to perform a large, appropriately powered randomized control trial to determine the effect of TLIP blocks on pain, physical function and disability, opioid consumption, and delirium in older adult undergoing spinal fusion.

ELIGIBILITY:
Inclusion Criteria:

* Are 65 or older
* Indicated for lumbar spinal fusion of less than or equal to 3 levels
* Undergoing elective surgery
* no contraindications to local anesthetic or procedures
* no severe cardiac or respiratory disease
* no preexisting cognitive dysfunction/dementia

Exclusion Criteria:

* 64 years old and younger
* emergency treatment
* pathologic fractures
* seeking revision surgery
* major liver or kidney dysfunction
* coexisting hematological disorder or irreversible abnormal coagulation
* patients with previous diagnosis of dementia or SLUMS score <20
* patient unable to communicate/cooperate/language barrier
* BMI>40
* allergy to study medications
* opioid tolerant (oral opioid intake morphine equivalent =< 60 mg/day)
* other sources of chronic pain like fibromyalgia
* patients with associated significant CNS or respiratory disease (home oxygen requirements)
* incarcerated patients
* psychiatric illnesses preoperative neurological deficits greater than one motor group, less than three out of five motor functions
* pregnant or breast feeding

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Score | Change assessed from pre-surgery to 12 weeks post-operatively.
  Change in pain will be assessed using the Numerical Rating Score Questionnaire immediately before surgery and at 2, 6 and 12 weeks post-operatively.
Daily Pain Trajectory | Change assessed from 1 day to 30 days post-operatively
  Change in pain will be assessed using the Daily Pain Trajectory survey each day post-operatively for 30 days.
Pain Catastrophizing | Change from Pre-operation score to 12 weeks post-operatively
  Change in pain catastrophizing and severity will be assessed using the Pain Catastrophizing scale immediately before surgery and at 2, 6, and 12 weeks post-operatively.
Pain Fear and Avoidance | Change from Pre-operation score to 12 weeks post-operatively
  Change in pain fear and subject avoidance will be assessed using the Pain Fear and Avoidance Questionnaire immediately before surgery and at 2, 6, and 12 weeks post-operatively.
Pain Interference | Change from Pre-operation score to 12 weeks post-operatively
  Change in how pain interferes with patient physical, emotional, and social functioning will be assessed using the PROMIS - Pain Interference questionnaire immediately before surgery and at 2, 6, and 12 weeks post-operatively.
Generalized Anxiety Disorder | Change from pre-operation score to 12 weeks post-operatively
  Change in severity measurement of generalized anxiety disorder assessed using the Generalized Anxiety Disorder 7 item scale immediately before surgery and at 2, 6, and 12 weeks post-operatively.
Personal Health Questionnaire Depression Scale | Change from pre-operation score to 12 weeks post-operatively
  Change in depression will be assessed using the Personal Health Questionnaire Depression Scale measured immediately before surgery and at 2, 6, and 12 weeks post-operatively.
Oswestry disability index | Change from Pre-operative score to 12 weeks post-operatively
  Change in disability score will be assessed using the Oswestry disability index measured immediately before surgery and at 2, 6, and 12 weeks post-operatively.
Tampa Scale of Kinesiophobia | Change from Pre-operative score to 12 weeks post-operatively
  Change in kinesiophobia will be assessed using the Tampa Scale of Kinesiophobia measured immediately before surgery and at 2, 6, and 12 weeks post-operatively.
Delirium Rating Scale-Revised-98 | Change from Pre-operative score to 12 weeks post-operatively
  Change in delirium severity will be assessed using the Delirium Rating Scale-Revised-98 16 item clinician rated scale measured immediately before surgery and at 1 day, 2 days, 3 days, 2 weeks, 6 weeks, and 12 weeks post-operatively.
3D-CAM-S and 3D-CAM-ICU | Change from Pre-operative score to 12 weeks post-operatively
  Change in delirium symptoms will be assessed using the 3D-CAM-S and 3D-CAM-ICU Questionnaire measured immediately before surgery and at 1 day, 2 days, 3 days, 2 weeks, 6 weeks, and 12 weeks post-operatively.
Modified Telephone Interview of Cognitive Status | Change from Pre-operative score to 12 weeks post-operatively
  Change in cognitive status will be assessed using the Modified Telephone Interview of cognitive Status measured immediately before surgery and at 6, and 12 weeks post-operatively.
Saint Louis University Mental Status Examination (SLUMs) | Change from Pre-operative score to 12 weeks post-operatively.
  Change in baseline cognition will be assessed using the Saint Louis University Mental Status Examination measured immediately before surgery and at 2, 6, and 12 weeks post-operatively.

SECONDARY OUTCOMES:
Opioid Use | Change from pre-operative score through 12 weeks post-operatively
  Opioid use will be calculated pre- and post-operatively using the Morphine Milligram Equivalents from patient self-reports.
Opioid Side Effects and Likability Questionnaire | Change from 1 week post-operative results to 4 weeks post-operation.
  Change in adverse events related to opioid side effects and complications will be assessed using the Opioid Side Effects and Likeability Questionnaire measured 1 week and 4 weeks post-operatively.
Self-reported Adverse Events | Change from pre-operative result through 12 weeks post-operatively.
  Change in adverse events related to opioid use and post-surgical outcomes will be collected post-operatively through the electronic health record from patient self-report. This will be measured immediately before surgery and 1, 2, 4, 6, and 12 weeks post-operatively
Length of Hospitalization | Through study completion, 16 months
  The length of time patients were hospitalized will be collected through the electronic health record.
Disposition to skilled-facilities | Through study completion, 16 months
  Where patients are dispositioned post-operatively will be collected through the electronic health record.
90-day Readmission Rates | Through study completion, 16 months
  The 90-day readmission rates will be collected through the electronic health record.
Blood test for Inflammation | Measured Immediately before surgery and 1 day post-operatively
  Blood test for IL-10, MCP-1, NfL, IL-6, and IL-8 will be done pre- and post-surgery for presence and levels of IL-10, MCP-1, NfL, IL-6, and IL-8.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine R Olinger, MD, Principal Investigator — Clinical Assistant Professor
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brown CH 4th, LaFlam A, Max L, Wyrobek J, Neufeld KJ, Kebaish KM, Cohen DB, Walston JD, Hogue CW, Riley LH. Delirium After Spine Surgery in Older Adults: Incidence, Risk Factors, and Outcomes. J Am Geriatr Soc. 2016 Oct;64(10):2101-2108. doi: 10.1111/jgs.14434. Epub 2016 Oct 3. PMID 27696373
- [Background] Lynch EP, Lazor MA, Gellis JE, Orav J, Goldman L, Marcantonio ER. The impact of postoperative pain on the development of postoperative delirium. Anesth Analg. 1998 Apr;86(4):781-5. doi: 10.1097/00000539-199804000-00019. PMID 9539601
- [Background] Morrison RS, Magaziner J, Gilbert M, Koval KJ, McLaughlin MA, Orosz G, Strauss E, Siu AL. Relationship between pain and opioid analgesics on the development of delirium following hip fracture. J Gerontol A Biol Sci Med Sci. 2003 Jan;58(1):76-81. doi: 10.1093/gerona/58.1.m76. PMID 12560416
- [Background] Wenk M, Liljenqvist U, Kaulingfrecks T, Gurlit S, Ermert T, Popping DM, Mollmann M. Intra- versus postoperative initiation of pain control via a thoracic epidural catheter for lumbar spinal fusion surgery. Minerva Anestesiol. 2018 Jul;84(7):796-802. doi: 10.23736/S0375-9393.17.12136-X. Epub 2017 Oct 4. PMID 28984097
- [Background] Chen K, Wang L, Ning M, Dou L, Li W, Li Y. Evaluation of ultrasound-guided lateral thoracolumbar interfascial plane block for postoperative analgesia in lumbar spine fusion surgery: a prospective, randomized, and controlled clinical trial. PeerJ. 2019 Oct 28;7:e7967. doi: 10.7717/peerj.7967. eCollection 2019. PMID 31681518
- [Background] Ye Y, Bi Y, Ma J, Liu B. Thoracolumbar interfascial plane block for postoperative analgesia in spine surgery: A systematic review and meta-analysis. PLoS One. 2021 May 21;16(5):e0251980. doi: 10.1371/journal.pone.0251980. eCollection 2021. PMID 34019598
- [Background] Deyo RA, Weinstein JN. Low back pain. N Engl J Med. 2001 Feb 1;344(5):363-70. doi: 10.1056/NEJM200102013440508. No abstract available. PMID 11172169
- [Background] Cassidy JD, Carroll LJ, Cote P. The Saskatchewan health and back pain survey. The prevalence of low back pain and related disability in Saskatchewan adults. Spine (Phila Pa 1976). 1998 Sep 1;23(17):1860-6; discussion 1867. doi: 10.1097/00007632-199809010-00012. PMID 9762743
- [Background] Khalifeh JM, Dibble CF, Hawasli AH, Ray WZ. Patient-Reported Outcomes Measurement Information System physical function and pain interference in spine surgery. J Neurosurg Spine. 2019 Apr 26;31(2):165-174. doi: 10.3171/2019.2.SPINE181237. Print 2019 Aug 1. PMID 31026819
- [Background] Khanna AK, Bergese SD, Jungquist CR, Morimatsu H, Uezono S, Lee S, Ti LK, Urman RD, McIntyre R Jr, Tornero C, Dahan A, Saager L, Weingarten TN, Wittmann M, Auckley D, Brazzi L, Le Guen M, Soto R, Schramm F, Ayad S, Kaw R, Di Stefano P, Sessler DI, Uribe A, Moll V, Dempsey SJ, Buhre W, Overdyk FJ; PRediction of Opioid-induced respiratory Depression In patients monitored by capnoGraphY (PRODIGY) Group Collaborators. Prediction of Opioid-Induced Respiratory Depression on Inpatient Wards Using Continuous Capnography and Oximetry: An International Prospective, Observational Trial. Anesth Analg. 2020 Oct;131(4):1012-1024. doi: 10.1213/ANE.0000000000004788. PMID 32925318
- [Background] Vila H Jr, Smith RA, Augustyniak MJ, Nagi PA, Soto RG, Ross TW, Cantor AB, Strickland JM, Miguel RV. The efficacy and safety of pain management before and after implementation of hospital-wide pain management standards: is patient safety compromised by treatment based solely on numerical pain ratings? Anesth Analg. 2005 Aug;101(2):474-480. doi: 10.1213/01.ANE.0000155970.45321.A8. PMID 16037164
- [Background] Rakel BA, Zimmerman BM, Geasland K, Embree J, Clark CR, Noiseux NO, Callaghan JJ, Herr K, Walsh D, Sluka KA. Transcutaneous electrical nerve stimulation for the control of pain during rehabilitation after total knee arthroplasty: A randomized, blinded, placebo-controlled trial. Pain. 2014 Dec;155(12):2599-2611. doi: 10.1016/j.pain.2014.09.025. Epub 2014 Sep 28. PMID 25270585
- [Background] Coronado RA, George SZ, Devin CJ, Wegener ST, Archer KR. Pain Sensitivity and Pain Catastrophizing Are Associated With Persistent Pain and Disability After Lumbar Spine Surgery. Arch Phys Med Rehabil. 2015 Oct;96(10):1763-70. doi: 10.1016/j.apmr.2015.06.003. Epub 2015 Jun 20. PMID 26101845
- [Background] Dunn LK, Durieux ME, Fernandez LG, Tsang S, Smith-Straesser EE, Jhaveri HF, Spanos SP, Thames MR, Spencer CD, Lloyd A, Stuart R, Ye F, Bray JP, Nemergut EC, Naik BI. Influence of catastrophizing, anxiety, and depression on in-hospital opioid consumption, pain, and quality of recovery after adult spine surgery. J Neurosurg Spine. 2018 Jan;28(1):119-126. doi: 10.3171/2017.5.SPINE1734. Epub 2017 Nov 10. PMID 29125426
- [Background] Nwankwo VC, Jiranek WA, Green CL, Allen KD, George SZ, Bettger JP. Resilience and pain catastrophizing among patients with total knee arthroplasty: a cohort study to examine psychological constructs as predictors of post-operative outcomes. Health Qual Life Outcomes. 2021 May 1;19(1):136. doi: 10.1186/s12955-021-01772-2. PMID 33933091
- [Background] Sanders RD, Pandharipande PP, Davidson AJ, Ma D, Maze M. Anticipating and managing postoperative delirium and cognitive decline in adults. BMJ. 2011 Jul 20;343:d4331. doi: 10.1136/bmj.d4331. No abstract available. PMID 21775401
- [Background] Ely EW, Gautam S, Margolin R, Francis J, May L, Speroff T, Truman B, Dittus R, Bernard R, Inouye SK. The impact of delirium in the intensive care unit on hospital length of stay. Intensive Care Med. 2001 Dec;27(12):1892-900. doi: 10.1007/s00134-001-1132-2. Epub 2001 Nov 8. PMID 11797025
- [Background] Mason SE, Noel-Storr A, Ritchie CW. The impact of general and regional anesthesia on the incidence of post-operative cognitive dysfunction and post-operative delirium: a systematic review with meta-analysis. J Alzheimers Dis. 2010;22 Suppl 3:67-79. doi: 10.3233/JAD-2010-101086. PMID 20858956
- [Background] Fong HK, Sands LP, Leung JM. The role of postoperative analgesia in delirium and cognitive decline in elderly patients: a systematic review. Anesth Analg. 2006 Apr;102(4):1255-66. doi: 10.1213/01.ane.0000198602.29716.53. PMID 16551934
- [Background] Leung JM, Sands LP, Lim E, Tsai TL, Kinjo S. Does preoperative risk for delirium moderate the effects of postoperative pain and opiate use on postoperative delirium? Am J Geriatr Psychiatry. 2013 Oct;21(10):946-56. doi: 10.1016/j.jagp.2013.01.069. Epub 2013 May 6. PMID 23659900
- [Background] Vaurio LE, Sands LP, Wang Y, Mullen EA, Leung JM. Postoperative delirium: the importance of pain and pain management. Anesth Analg. 2006 Apr;102(4):1267-73. doi: 10.1213/01.ane.0000199156.59226.af. PMID 16551935
- [Background] Berger M, Terrando N, Smith SK, Browndyke JN, Newman MF, Mathew JP. Neurocognitive Function after Cardiac Surgery: From Phenotypes to Mechanisms. Anesthesiology. 2018 Oct;129(4):829-851. doi: 10.1097/ALN.0000000000002194. PMID 29621031
- [Background] Hand WR, Taylor JM, Harvey NR, Epperson TI, Gunselman RJ, Bolin ED, Whiteley J. Thoracolumbar interfascial plane (TLIP) block: a pilot study in volunteers. Can J Anaesth. 2015 Nov;62(11):1196-200. doi: 10.1007/s12630-015-0431-y. Epub 2015 Jul 7. PMID 26149600
- [Background] Garg B, Ahuja K, Khanna P, Sharan AD. Regional Anesthesia for Spine Surgery. Clin Spine Surg. 2021 Jun 1;34(5):163-170. doi: 10.1097/BSD.0000000000001096. Epub 2020 Oct 9. PMID 33044273
- [Background] Bicak M, Aktas U, Salik F, Akelma H, Bicak EA, Kaya S. Comparison of Thoracolumbar Interfascial Plane Block with the Application of Local Anesthesia in the Management of Postoperative Pain in Patients with Lumbar Disc Surgery. Turk Neurosurg. 2021;31(5):757-762. doi: 10.5137/1019-5149.JTN.33017-20.2. PMID 34374980
- [Background] Ueshima H, Hara E, Otake H. RETRACTED: Thoracolumbar interfascial plane block provides effective perioperative pain relief for patients undergoing lumbar spinal surgery; a prospective, randomized and double blinded trial. J Clin Anesth. 2019 Dec;58:12-17. doi: 10.1016/j.jclinane.2019.04.026. Epub 2019 Apr 25. PMID 31029989 (Retraction: PMID 35393187 J Clin Anesth. 2022 Aug;79:110690)
- [Background] Ohgoshi Y, Namiki R, Kori S, Matsukawa M. The use of ultrasound-guided thoracolumbar interfascial plane block for multi-level lumbar spinal surgery. J Clin Anesth. 2017 Feb;37:162. doi: 10.1016/j.jclinane.2016.12.025. Epub 2017 Jan 10. No abstract available. PMID 28235513
- [Background] Tseng V, Xu JL. Erector Spinae Plane Block for Postoperative Analgesia in Lumbar Spine Surgery: Is There a Better Option? J Neurosurg Anesthesiol. 2021 Jan;33(1):92. doi: 10.1097/ANA.0000000000000631. No abstract available. PMID 31343504
- [Background] Ueshima H. Retraction notice to "Lumbar thoracolumbar interfascial plane block provides effective analgesia for spondylosis" [J. Clin. Anesth. 57 (2019)37]. J Clin Anesth. 2022 Aug;79:110762. doi: 10.1016/j.jclinane.2022.110762. Epub 2022 Apr 4. No abstract available. PMID 35393185
- [Background] Morgenstern C, Ramirez-Paesano C, Juanola Galceran A, Morgenstern R. Thoracolumbar Interfascial Plane Block Results in Opioid-Free Postoperative Recovery After Percutaneous/Endoscopic Transforaminal Lumbar Interbody Fusion Surgery. World Neurosurg. 2021 Sep;153:e473-e480. doi: 10.1016/j.wneu.2021.06.152. Epub 2021 Jul 6. PMID 34242827
- [Background] Gao H, Ma HJ, Li YJ, Yin C, Li Z. Prevalence and risk factors of postoperative delirium after spinal surgery: a meta-analysis. J Orthop Surg Res. 2020 Apr 9;15(1):138. doi: 10.1186/s13018-020-01651-4. PMID 32272939
- [Background] Farag E, Seif J. Thoracolumbar interfascial block (TLIP): A new technique of interfascial plane blocks. J Clin Anesth. 2020 May;61:109640. doi: 10.1016/j.jclinane.2019.109640. Epub 2019 Oct 28. No abstract available. PMID 31672416
- [Background] Shin C, Lee SH, Han KM, Yoon HK, Han C. Comparison of the Usefulness of the PHQ-8 and PHQ-9 for Screening for Major Depressive Disorder: Analysis of Psychiatric Outpatient Data. Psychiatry Investig. 2019 Apr;16(4):300-305. doi: 10.30773/pi.2019.02.01. Epub 2019 Apr 24. PMID 31042692
- [Background] Von Korff M, Saunders K, Thomas Ray G, Boudreau D, Campbell C, Merrill J, Sullivan MD, Rutter CM, Silverberg MJ, Banta-Green C, Weisner C. De facto long-term opioid therapy for noncancer pain. Clin J Pain. 2008 Jul-Aug;24(6):521-7. doi: 10.1097/AJP.0b013e318169d03b. PMID 18574361
- [Background] Ahn SH, Choi JH, Im CS, Kim TS, Kim JL. A Comparison of the Severe Cognitive Impairment Rating Scale With the Mini-Mental State Examination and Delirium Rating Scale-Revised-98 for Delirium: A Cross-sectional Study. Psychosomatics. 2017 Nov-Dec;58(6):643-651. doi: 10.1016/j.psym.2017.08.002. Epub 2017 Aug 5. PMID 29032807
- [Background] Marcantonio ER, Ngo LH, O'Connor M, Jones RN, Crane PK, Metzger ED, Inouye SK. 3D-CAM: derivation and validation of a 3-minute diagnostic interview for CAM-defined delirium: a cross-sectional diagnostic test study. Ann Intern Med. 2014 Oct 21;161(8):554-61. doi: 10.7326/M14-0865. PMID 25329203
- [Background] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446
- [Background] Olbert M, Eckert S, Morgeli R, Kruppa J, Spies CD. Validation of 3-minute diagnostic interview for CAM-defined Delirium to detect postoperative delirium in the recovery room: A prospective diagnostic study. Eur J Anaesthesiol. 2019 Sep;36(9):683-687. doi: 10.1097/EJA.0000000000001048. PMID 31306183
- [Background] Tariq SH, Tumosa N, Chibnall JT, Perry MH 3rd, Morley JE. Comparison of the Saint Louis University mental status examination and the mini-mental state examination for detecting dementia and mild neurocognitive disorder--a pilot study. Am J Geriatr Psychiatry. 2006 Nov;14(11):900-10. doi: 10.1097/01.JGP.0000221510.33817.86. PMID 17068312
- [Background] Yadeau JT, Liu SS, Rade MC, Marcello D, Liguori GA. Performance characteristics and validation of the Opioid-Related Symptom Distress Scale for evaluation of analgesic side effects after orthopedic surgery. Anesth Analg. 2011 Aug;113(2):369-77. doi: 10.1213/ANE.0b013e31821ae3f7. Epub 2011 Apr 27. PMID 21525182
- [Background] Jamison RN, Dorado K, Mei A, Edwards RR, Martel MO. Influence of opioid-related side effects on disability, mood, and opioid misuse risk among patients with chronic pain in primary care. Pain Rep. 2017 Mar 6;2(2):e589. doi: 10.1097/PR9.0000000000000589. eCollection 2017 Mar. PMID 29392205
- [Background] Glare P, Walsh D, Sheehan D. The adverse effects of morphine: a prospective survey of common symptoms during repeated dosing for chronic cancer pain. Am J Hosp Palliat Care. 2006 Jun-Jul;23(3):229-35. doi: 10.1177/1049909106289068. PMID 17060284
- [Background] Dailey DL, Vance CGT, Rakel BA, Zimmerman MB, Embree J, Merriwether EN, Geasland KM, Chimenti R, Williams JM, Golchha M, Crofford LJ, Sluka KA. Transcutaneous Electrical Nerve Stimulation Reduces Movement-Evoked Pain and Fatigue: A Randomized, Controlled Trial. Arthritis Rheumatol. 2020 May;72(5):824-836. doi: 10.1002/art.41170. Epub 2020 Mar 18. PMID 31738014
- [Background] Driban JB, Morgan N, Price LL, Cook KF, Wang C. Patient-Reported Outcomes Measurement Information System (PROMIS) instruments among individuals with symptomatic knee osteoarthritis: a cross-sectional study of floor/ceiling effects and construct validity. BMC Musculoskelet Disord. 2015 Sep 14;16:253. doi: 10.1186/s12891-015-0715-y. PMID 26369412
- [Background] Quan H, Li B, Couris CM, Fushimi K, Graham P, Hider P, Januel JM, Sundararajan V. Updating and validating the Charlson comorbidity index and score for risk adjustment in hospital discharge abstracts using data from 6 countries. Am J Epidemiol. 2011 Mar 15;173(6):676-82. doi: 10.1093/aje/kwq433. Epub 2011 Feb 17. PMID 21330339
- [Background] Sim J, Lewis M. The size of a pilot study for a clinical trial should be calculated in relation to considerations of precision and efficiency. J Clin Epidemiol. 2012 Mar;65(3):301-8. doi: 10.1016/j.jclinepi.2011.07.011. Epub 2011 Dec 9. PMID 22169081
- [Background] Asher AL, Kerezoudis P, Mummaneni PV, Bisson EF, Glassman SD, Foley KT, Slotkin JR, Potts EA, Shaffrey ME, Shaffrey CI, Coric D, Knightly JJ, Park P, Fu KM, Devin CJ, Archer KR, Chotai S, Chan AK, Virk MS, Bydon M. Defining the minimum clinically important difference for grade I degenerative lumbar spondylolisthesis: insights from the Quality Outcomes Database. Neurosurg Focus. 2018 Jan;44(1):E2. doi: 10.3171/2017.10.FOCUS17554. PMID 29290132
- [Background] Goudman L, Smedt A, Forget P, Moens M. Determining the Minimal Clinical Important Difference for Medication Quantification Scale III and Morphine Milligram Equivalents in Patients with Failed Back Surgery Syndrome. J Clin Med. 2020 Nov 21;9(11):3747. doi: 10.3390/jcm9113747. PMID 33233343
- [Background] Brock JL, Jain N, Phillips FM, Malik AT, Khan SN. Postoperative opioid cessation rates based on preoperative opioid use: analysis of common orthopaedic procedures. Bone Joint J. 2019 Dec;101-B(12):1570-1577. doi: 10.1302/0301-620X.101B12.BJJ-2019-0080.R2. PMID 31787005